CLINICAL TRIAL: NCT03049449
Title: Anti-CD30 CAR T Cells With Fully-human Binding Domains for Treating CD30-expressing Lymphomas Including Anaplastic Large Cell Lymphomas
Brief Title: T Cells Expressing a Fully-Human Anti-CD30 Chimeric Antigen Receptor for Treating CD30-Expressing Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Kochenderfer, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 170048; 17-C-0048
Record Dates: First submitted 2017-02-09; First posted 2017-02-10 (Actual); Results first posted 2022-05-25 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Lymphoma, Large-Cell, Anaplastic; Enteropathy-Associated T-Cell Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Extranodal NK-T-Cell; Lymphoma, T-Cell, Peripheral
Keywords: Gray Zone Lymphoma; Immunotherapy; Peripheral T-Cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Enteropathy-Associated T-Cell Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Extranodal NK-T-Cell; Lymphoma, T-Cell, Peripheral; Immunoblastic Lymphadenopathy | interventions — Ki-1 Antigen; Receptors, Chimeric Antigen; Automobiles; Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chimeric Antigen Receptor (CAR)+ T cells (Experimental): All patients will be receiving starting dose: 0.3x10^6 Chimeric Antigen Receptor (CAR)+ T cells/kg (weight based dosing) (up to a maximum dose of 18x10^6 CAR+ T cells/kg) infuse on day 0 and Cyclophosphamide: 300 or 500 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 and Fludarabine: 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
  Interventions: Biological: Anti-Tumor Necrosis Factor (TNF) Receptor Superfamily Member 8 (CD30) Chimeric Antigen Receptor (CAR) T cells; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: Anti-Tumor Necrosis Factor (TNF) Receptor Superfamily Member 8 (CD30) Chimeric Antigen Receptor (CAR) T cells — Dose-escalation trial starting dose: 0.3x10^6 Chimeric Antigen Receptor (CAR)+ T cells/kg (weight based dosing) (up to a maximum dose of 18x10^6 CAR+ T cells/kg) infuse on day 0
Drug: Cyclophosphamide — 300 or 500 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3
  Other Names: Cytoxan
Drug: Fludarabine — 30 mg/m^2 intravenous (IV) infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
  Other Names: Fludara

SUMMARY:
Background:

* Improved treatments for a variety of treatment-resistant, TNFRSF8 (CD30)-expressing malignancies including Hodgkin lymphoma, anaplastic large cell lymphoma, and other CD30- expressing lymphomas are needed.
* T cells can be genetically modified to express chimeric antigen receptors (CARs) that specifically target malignancy-associated antigens.
* Autologous T cells genetically modified to express CARs targeting the B-cell antigen B-lymphocyte antigen CD19 (CD19) have caused complete remissions in a small number of patients with lymphoma. These results demonstrate that CAR-expressing T cells can have anti-lymphoma activity in humans.
* CD30 expression can be easily detected by immunohistochemistry on lymphoma cells, which allows selection of CD30-expressing malignancies for treatment.
* CD30 is not known to be expressed by normal cells except for a small number of activated lymphocytes.
* We have constructed a novel fully-human anti-CD30 CAR that can specifically recognize CD30-expressing target cells in vitro and eradicate CD30-expressing tumors in mice.
* This particular CAR has not been tested before in humans.
* Possible toxicities include cytokine-associated toxicities such as fever, hypotension, and neurological toxicities. Elimination of a small number of normal activated lymphocytes is possible, and unknown toxicities are also possible.

Objectives:

Primary

-Determine the safety and feasibility of administering T-cells expressing a novel fully human anti-CD30 CAR to patients with advanced CD30-expressing lymphomas.

Eligibility:

* Patients must have anaplastic large cell lymphoma, peripheral T-cell lymphoma not otherwise specified, diffuse large B-cell lymphoma not otherwise specified, primary mediastinal B-cell lymphoma, grey zone lymphoma, enteropathy associated T-cell lymphoma, or extranodal natural killer (NK)/T-cell lymphoma, nasal type
* Patients must have malignancy that is both measurable on a computed tomography (CT) scan with a largest diameter of at least 1.5 cm and possessing increased metabolic activity detectable by positron emission tomography (PET) scan. Alternatively, patients with lymphoma detected by flow cytometry of bone marrow are eligible.
* Patients must have a creatinine of 1.6 mg/dL or less and a normal cardiac ejection fraction.
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 is required.
* No active infections are allowed including evidence of active human immunodeficiency virus (HIV), hepatitis B, or hepatitis C. At the time of protocol enrollment patients must be seronegative for cytomegalovirus (CMV) by antibody testing or must have a negative blood CMV polymerase chain reaction (PCR).
* Absolute neutrophil count greater than or equal to 1000/micro L, platelet count greater than or equal to 55,000/micro L, hemoglobin greater than or equal to 8g/dL
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less or equal to 3 times the upper limit of the institutional normal unless liver involvement by malignancy is demonstrated.
* At least 14 days must elapse between the time of any prior systemic treatment (including corticosteroids above 5 mg/day of prednisone or equivalent corticosteroid dose) and initiation of required leukapheresis.
* Clear CD30 expression must be detected on 75% or more of malignant cells from either bone marrow or lymphoma mass by flow cytometry or immunohistochemistry. The patient s malignancy will need to be assessed for CD30 expression by flow cytometry or immunohistochemistry performed at the National Institutes of Health (NIH). If unstained, paraffin-embedded bone marrow or lymphoma sections are available from prior biopsies, these can be used to determine CD30 expression by immunohistochemistry; otherwise, patients will need to come to the NIH for a biopsy to determine CD30 expression. The sample for CD30 expression can come from a biopsy obtained at any time before enrollment, unless the patient has received a prior anti-CD30 monoclonal antibody, in which case the sample must come from a biopsy following completion of the most recent anti-CD30 monoclonal antibody treatment.
* Eligible patients with diffuse large B-cell lymphoma or primary mediastinal B-cell lymphoma must have received 2 prior treatment regimens at least 1 of which included an anthracycline and an anti-CD20 monoclonal antibody.
* Patients who have never had an allogeneic hematopoietic stem cell transplant as well as patients who have had a 9/10 or 10/10 human leukocyte antigen (HLA)-matched sibling or a 9/10 or 10/10 HLA- matched unrelated donor hematopoietic stem cell transplant are potentially eligible.
* Women who are pregnant or plan to become pregnant will be excluded.

DETAILED DESCRIPTION:
Background:

* Improved treatments for a variety of treatment-resistant, TNFRSF8 (CD30)-expressing malignancies including Hodgkin lymphoma, anaplastic large cell lymphoma, and other CD30- expressing lymphomas are needed.
* T cells can be genetically modified to express chimeric antigen receptors (CARs) that specifically target malignancy-associated antigens.
* Autologous T cells genetically modified to express CARs targeting the B-cell antigen B-lymphocyte antigen CD19 (CD19) have caused complete remissions in a small number of patients with lymphoma. These results demonstrate that CAR-expressing T cells can have anti-lymphoma activity in humans.
* CD30 expression can be easily detected by immunohistochemistry on lymphoma cells, which allows selection of CD30-expressing malignancies for treatment.
* CD30 is not known to be expressed by normal cells except for a small number of activated lymphocytes.
* We have constructed a novel fully-human anti-CD30 CAR that can specifically recognize CD30-expressing target cells in vitro and eradicate CD30-expressing tumors in mice.
* This particular CAR has not been tested before in humans.
* Possible toxicities include cytokine-associated toxicities such as fever, hypotension, and neurological toxicities. Elimination of a small number of normal activated lymphocytes is possible, and unknown toxicities are also possible.

Objectives:

Primary

-Determine the safety and feasibility of administering T-cells expressing a novel fully-human anti-CD30 CAR to patients with advanced CD30-expressing lymphomas.

Eligibility:

* Patients must have anaplastic large cell lymphoma, angioimmunoblastic T-cell lymphoma, peripheral T-cell lymphoma not otherwise specified, diffuse large B-cell lymphoma not otherwise specified, primary mediastinal B-cell lymphoma, grey zone lymphoma, enteropathy-associated T-cell lymphoma, or extranodal natural killer (NK)//T-cell lymphoma, nasal type
* Patients must have malignancy that is both measurable on a computed tomography (CT) scan with a largest diameter of at least 1.5 cm and possessing increased metabolic activity detectable by positron emission tomography (PET) scan. Alternatively, patients with lymphoma detected by flow cytometry of bone marrow are eligible.
* Patients must have a creatinine of 1.6 mg/dL or less and a normal cardiac ejection fraction.
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 is required.
* No active infections are allowed including evidence of active human immunodeficiency virus (HIV), hepatitis B, or hepatitis C. At the time of protocol enrollment, patients must be seronegative for cytomegalovirus (CMV) by antibody testing or must have a negative blood CMV polymerase chain reaction (PCR).
* Absolute neutrophil count greater than or equal to 1000/micro L, platelet count greater than or equal to 55,000/micro L, hemoglobin greater than or equal to 8g/dL
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less or equal to 3 times the upper limit of the institutional normal unless liver involvement by malignancy is demonstrated.
* At least 14 days must elapse between the time of any prior systemic treatment (including corticosteroids above 5 mg/day of prednisone or equivalent corticosteroid dose) and initiation of required leukapheresis.
* Clear CD30 expression must be detected on 75% or more of malignant cells from either bone marrow or lymphoma mass by flow cytometry or immunohistochemistry. The patient s malignancy will need to be assessed for CD30 expression by flow cytometry or immunohistochemistry performed at the National Institutes of Health (NIH). If unstained, paraffin-embedded bone marrow or lymphoma sections are available from prior biopsies, these can be used to determine CD30 expression by immunohistochemistry; otherwise, patients will need to come to the NIH for a biopsy to determine CD30 expression. The sample for CD30 expression can come from a biopsy obtained at any time before enrollment, unless the patient has received a prior anti-CD30 monoclonal antibody, in which case the sample must come from a biopsy following completion of the most recent anti-CD30 monoclonal antibody treatment.
* Eligible patients with diffuse large B-cell lymphoma or primary mediastinal B-cell lymphoma must have received 2 prior treatment regimens at least 1 of which included an anthracycline and an anti-CD20 monoclonal antibody.
* Patients who have never had an allogeneic hematopoietic stem cell transplant as well as patients who have had a 9/10 or 10/10 human leukocyte antigen (HLA)-matched sibling or a 9/10 or 10/10 HLA- matched unrelated donor hematopoietic stem cell transplant are potentially eligible.
* Women who are pregnant or plan to become pregnant will be excluded.

Design:

* This is a phase I dose-escalation trial.
* Patients will undergo leukapheresis.
* T cells obtained by leukapheresis will be genetically modified to express an anti-CD30 CAR.
* Patients will receive a lymphocyte-depleting chemotherapy conditioning regimen with the intent of enhancing the activity of the infused anti-CD30 CAR-expressing T cells.
* A chemotherapy conditioning regimen of cyclophosphamide and fludarabine will be administered prior to all CAR T-Cell infusions. Fludarabine will be given on the same days as the cyclophosphamide.
* Two days after the chemotherapy ends, patients will receive an infusion of anti-CD30-CAR-expressing T cells.
* The initial dose level of this dose-escalation trial will be 0.3x10(6) CAR+ T cells/kg of recipient bodyweight for Cohort 1. The initial dose level will be 1 x 10 (6) CAR+T cells/kg for Cohort 2.
* The cell dose administered will be escalated until a maximum tolerated dose is determined.
* Following the T-cell infusion, there is a mandatory 9-day inpatient hospitalization to monitor for toxicity.
* Outpatient follow-up is planned for 2 weeks and 1, 2, 3, 4, 6, 9, and 12 months after the CAR T-cell infusion. Long-term gene-therapy follow-up consisting of yearly visits to a doctor near the patients home for 4 more years and then yearly telephone contact for 10 additional years will be required.
* As of Amendment E (Protocol version: 08/03/2018), repeat treatments consisting of the conditioning chemotherapy followed by a CAR T-cell infusion at the maximum tolerated dose (MTD) for the patients cohort are allowed for eligible patients with any best responses except continuing complete remission or progressive malignancy.
* Re-enrollment will be allowed for a small number of subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

Malignancy Criteria:

* Patients must have anaplastic large cell lymphoma, angioimmunoblastic T-cell lymphoma, peripheral T-cell lymphoma not otherwise specified, diffuse large B-cell lymphoma not otherwise specified, primary mediastinal B-cell lymphoma, grey zone lymphoma, enteropathy-associated T-cell lymphoma, or extranodal natural killer (NK)/T-cell lymphoma, nasal type
* Clear TNFRSF8 (CD30) expression must be detected on 75% or more of malignant cells from either bone marrow or lymphoma mass by flow cytometry or immunohistochemistry. The patient's malignancy will need to be assessed for CD30 expression by flow cytometry or immunohistochemistry performed at the National Institutes of Health (NIH). If unstained, paraffin-embedded bone marrow or lymphoma sections are available from prior biopsies, these can be used to determine CD30 expression by immunohistochemistry; otherwise, patients will need to come to the NIH for a biopsy to determine CD30 expression. The sample for CD30 expression can come from a biopsy obtained at any time before enrollment, unless the patient has received a prior anti-CD30 monoclonal antibody, in which case the sample must come from a biopsy following completion of the most recent anti-CD30 monoclonal antibody treatment.
* Eligible patients with diffuse large B-cell lymphoma or primary mediastinal B-cell lymphoma must have received 2 prior treatment regimens at least 1 of which included an anthracycline and an anti-B-lymphocyte antigen CD20 (CD20) monoclonal antibody.
* Patients must have measurable malignancy as defined by at least one of the criteria below.
* Lymphoma mass that is measurable (minimum 1.5 cm in largest diameter) by computed tomography (CT) scan is required unless bone marrow lymphoma is detectable.
* For a lymphoma mass to count as measurable malignancy, it must have abnormally increased metabolic activity when assessed by positron emission tomography (PET) scan.
* For lymphoma with only bone marrow involvement, no mass is necessary, but if a mass is not present, bone marrow malignancy must be detectable by flow cytometry.

Other Inclusion Criteria:

* Greater than or equal to 18 years of age and less than or equal to age 73.
* Able to understand and sign the Informed Consent Document.
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0-2
* Room air oxygen saturation of 92% or greater
* Male patients and must be willing to practice birth control from the time of enrollment on this study and for four months following the final CAR T-cell infusion. Pre-menopausal patients (female patients who have had a menstrual period within the last year) must be willing to practice birth control from the time of enrollment and for one year following the final CAR T cell infusion.
* Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune -competence and thus are less responsive to the experimental treatment and more susceptible to its toxicities.)
* Seronegative for Human T-cell lymphotropic virus type 1 (HTLV-1).
* Negative for hepatitis B surface antigen. Positive hepatitis B tests can be further evaluated by confirmatory tests; and if confirmatory tests are negative, the patient can be enrolled.
* Seronegative for hepatitis C antibody unless antigen negative. If hepatitis C antibody test is positive, then patients must be tested for the presence of ribonucleic acid (RNA) by Reverse transcription polymerase chain reaction (RT-PCR) and be Hepatitis C (HCV) RNA negative to be enrolled.
* A patient with a prior history of hepatitis B or a prior history of hepatitis C may participate, as long as the patient s viral hepatitis has been treated, and the patient has no detectable Hepatitis B (HBV) deoxyribonucleic acid (DNA) or HCV RNA.
* At time of protocol enrollment, the patient should be negative for cytomegalovirus (CMV) by antibody testing or by PCR. In case of disagreement between these 2 CMV tests, the tests will be repeated, and Dept. of Laboratory Medicine consulted.
* Absolute neutrophil count greater than or equal to 1000/mm^3 without the support of filgrastim or other growth factors.
* Platelet count greater than or equal to 55,000/mm^3
* Hemoglobin greater than 8.0 g/dl. Transfusion support is allowed.
* Less than 5% malignant cells in the peripheral blood leukocytes
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less or equal to 3 times the upper limit of the institutional normal unless liver involvement by malignancy is demonstrated.
* Serum creatinine less than or equal to 1.6 mg/dL.
* Total bilirubin less than or equal to 2.0 mg/dl.
* At least 14 days must have elapsed since any prior systemic therapy prior to apheresis and prior to the initiation of chemotherapy (including systemic corticosteroids at doses greater than prednisone 5 mg/day or the equivalent corticosteroid doses). Because this protocol requires collection of autologous blood cells by leukapheresis in order to prepare CAR T cells, systemic anti-malignancy therapy including systemic corticosteroid therapy at doses greater than prednisone 5 mg/day or the equivalent corticosteroid doses is not allowed within 14 days prior to the required leukapheresis. NOTE: Because of the long half-life and potential to affect CAR T-cells, 30 days must elapse from the time of administration of anti-Programmed cell death protein 1 (PD-1) or anti-Programmed death-ligand 1 (PD-L1) antibodies or other agents that in the opinion of the PI can stimulate immune activity and infusion of CAR T-cells.
* Normal cardiac ejection fraction (greater than or equal to 50% by echocardiography) and no evidence of hemodynamically significant pericardial effusion as determined by an echocardiogram within 4 weeks of the start of the treatment protocol.
* Patients must not take corticosteroids at doses higher than 5 mg/day of prednisone or the equivalent for 14 days before apheresis, and for 14 days prior to the conditioning chemotherapy regimen.
* Patients must be willing to undergo endotracheal intubation, mechanical ventilation, dialysis, cardiopulmonary resuscitation (CPR), and electrical defibrillation. Patients must be willing to receive vasopressor drugs and all other standard intensive care unit interventions. Any living will must be amended to allow these interventions, or the patient will not eligible.
* Patients who have been treated on other protocols of genetically-modified T-cells at the National Institutes of Health (NIH) only are potentially eligible under these conditions:

  * At least 6 months have elapsed since the last genetically-modified T-cell therapy that the patient received and there is no evidence of replication-competent retroviruses (evidence must be provided from prior NIH gene-therapy protocol Principal Investigator) and persisting genetically-modified T cells are not detectable in the patient's blood (evidence must be provided by prior NIH gene-therapy protocol Principal Investigator).

Additional Inclusion Criteria Pertinent Only for Patients with Prior Allogeneic Transplantation:

* Recipients must have received an 9/10 or 10/10 HLA-matched sibling allogeneic hematopoietic stem cell transplant, or a 9/10 or 10/10 HLA-matched unrelated donor (URD) allo-HSCT for an eligible CD30+ lymphoma.
* Donor T cell engraftment after allo-Hematopoietic stem-cell transplantation (HSCT)(>90% donor chimerism of the T-cell compartment).
* Patients must be at least 90 days post-transplant.
* Patients must be off all systemic immunosuppressive drugs including corticosteroids at doses of greater than 5 mg/day prednisone or equivalent, if given for treatment of graft versus host disease, for at least 28 days prior to protocol enrollment and must remain off immunosuppressive drugs while enrolled on the protocol. Patients must not be taking any systemic steroids at doses greater than 5 mg/day prednisone or equivalent at all for 14 days prior to apheresis and initiation of chemotherapy. Topical corticosteroid preparations applied to the skin such as solutions, creams, and ointments are allowed. Inhaled corticosteroids are allowed, and corticosteroid eye drops are allowed.
* Prior donor lymphocyte infusions (DLIs) are not necessary.
* Either no evidence of graft versus host (GVHD) or minimal clinical evidence of acute GVHD and chronic GVHD while off of systemic immunosuppressive therapy for at least 28 days. Minimal clinical evidence of acute GVHD defined as grade 0 to I acute GVHD 109 Minimal evidence of chronic GVHD is defined as mild global score chronic GVHD (as defined by the 2005 NIH consensus project) or no chronic GVHD .107 Subjects with disease that is controlled to stage I acute GVHD or to mild global score chronic GVHD with local topical cutaneous steroids will be eligible for enrollment.

EXCLUSION CRITERIA:

* Patients with Hodgkin lymphoma are no longer eligible for participation (as of amendment G, Protocol version: 08/12/2019).
* Patients that require urgent therapy due to tumor mass effects or spinal cord compression.
* Patients with lymphoma masses 10.0 cm or larger in longest diameter will not be eligible.
* Patients that have active hemolytic anemia.
* Patients who are currently taking any medications for systemic anticoagulation other than aspirin will not be eligible.
* Patients with second malignancies in addition to their lymphoma are not eligible if the second malignancy has required treatment (including maintenance therapy) within the past 4 years or is not in complete remission. There are two exceptions to this criterion:

successfully treated non-metastatic basal cell or squamous cell skin carcinoma.

* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant. Women of child-bearing potential are defined as all women except women who are postmenopausal or who have had a hysterectomy. Postmenopausal will be defined as women over the age of 55 who have not had a menstrual period in at least 1 year.
* Active uncontrolled systemic infections (defined as infections causing fevers and infections requiring intravenous antibiotics when the intravenous antibiotics have been administered for less than 72 hours); active coagulation disorders or other major uncontrolled medical illnesses of the cardiovascular, respiratory, endocrine, renal, gastrointestinal, genitourinary or immune system; history of myocardial infarction; history of idiopathic ventricular tachycardia or ventricular fibrillation in the past 12 months or history of ventricular tachycardia or ventricular fibrillation (VT/VF) associated with VT/VF risk factors (e.g., QT prolongation and cardiomyopathy); active cardiac arrhythmias (Active atrial fibrillation is not allowed, but resolved atrial fibrillation is allowed.); active obstructive or restrictive pulmonary disease; or active autoimmune diseases such as rheumatoid arthritis.
* Patients will not be seen for screening appointments or enrolled on the protocol if they have been hospitalized within the 7 days prior to the screening appointment or the date of protocol enrollment.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease) , unless the immunodeficiency has been cured by allogeneic stem cell transplant.
* Systemic corticosteroid therapy at doses greater than 5 mg/day of prednisone or the equivalent dose is not allowed within 14 days prior to the required leukapheresis, or the initiation of the conditioning chemotherapy regimen. Corticosteroid creams, ointments, and eye drops are allowed.
* History of severe immediate hypersensitivity reaction to any of the agents used in this study.
* Patients with current central nervous system (CNS) involvement by malignancy (either by imaging or cerebrospinal fluid involvement or biopsy-proven).
* Patients currently taking anticoagulants.

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James N Kochenderfer, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share coded, linked data in an National Institutes of Health (NIH)-funded or approved public repository. Coded, linked data in Biomedical Translational Research Information System (BTRIS).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared before publication. And at the time of publication or shortly thereafter.
Access Criteria: An National Institutes of Health (NIH)-funded or approved public repository - Clinical Trials.gov, Biomedical Translational Research Information System (BTRIS), and publication and/or presentations.

REFERENCES:
- [Derived] Brudno JN, Natrakul DA, Karrs J, Patel N, Maass-Moreno R, Ahlman MA, Mikkilineni L, Mann J, Stroncek DF, Highfill SL, Fromm GC, Patel R, Pittaluga S, Kochenderfer JN. Transient responses and significant toxicities of anti-CD30 CAR T cells for CD30+ lymphomas: results of a phase 1 trial. Blood Adv. 2024 Feb 13;8(3):802-814. doi: 10.1182/bloodadvances.2023011470. PMID 37939262
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0048.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Escalation Cohort 1 Dose Level -1 - 0.15x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg: 0.15x10^6 Chimeric Antigen Receptor (CAR) T cells per kg of recipient bodyweight
  No participants were enrolled on dose level -1.
- Dose Escalation Cohort 1 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg: Participants who have not had an allogeneic hematopoietic stem cell transplant. 0.3x10^6 Chimeric Antigen Receptor (CAR) T cells per kg of recipient bodyweight
  Starting dose: 0.3x10^6 Chimeric Antigen Receptor (CAR)+ T cells/kg (weight based dosing) infuse on day 0 and Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 and Fludarabine: 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4,and -3
- Dose Escalation Cohort 1 Dose Level 2 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg: Participants who have not had an allogeneic hematopoietic stem cell transplant. 1.0x10^6 Chimeric Antigen Receptor (CAR) T cells per kg of recipient bodyweight
  1.0x10^6 Chimeric Antigen Receptor (CAR)+ T cells/kg (weight based dosing) infuse on day 0 and Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 and Fludarabine: 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
- Dose Escalation Cohort 1 Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg: Participants who have not had an allogeneic hematopoietic stem cell transplant. 3.0x10^6 Chimeric Antigen Receptor (CAR) T cells per kg of recipient bodyweight
  3.0x10^6 Chimeric Antigen Receptor (CAR)+ T cells/kg (weight based dosing) infuse on day 0 and Cyclophosphamide: This chemotherapy dose was changed part-way through the protocol, thus 4 participants received 500 mg/m^2 and 3 participants received 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 and Fludarabine: 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3.
- Dose Escalation Cohort 1 Dose Level 4 - 9.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg: Participants who have not had an allogeneic hematopoietic stem cell transplant. 9.0x10^6 Chimeric Antigen Receptor (CAR) T cells per kg of recipient bodyweight
  9.0 x10^6 Chimeric Antigen Receptor (CAR)+ T cells/kg (weight based dosing) infuse on day 0 and Cyclophosphamide: 500 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 and Fludarabine: 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
- Dose Escalation Cohort 1 Dose Level 5 - 18x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg: 18x10^6 Chimeric Antigen Receptor (CAR) T cells per kg of recipient bodyweight with a maximum dose of 216x10^7 CAR T cells.
  No participants were enrolled on dose level 5.
- Dose Escalation Cohort 2 Dose Level 1 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg: Participants who have had an Human Leukocyte Antigen (HLA)-matched sibling or an 8/8-HLA-matched unrelated donor transplant.
  1.0x10^6 Chimeric Antigen Receptor (CAR) T cells per kg of recipient bodyweight
  1.0 x10^6 Chimeric Antigen Receptor (CAR)+ T cells/kg (weight based dosing) infuse on day 0 and Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 and Fludarabine: 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
- Dose Escalation Cohort 2 Dose Level 2 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg: Participants who have had an Human Leukocyte Antigen (HLA)-matched sibling or an 8/8 HLA-matched unrelated donor transplant.
  3.0x10^6 Chimeric Antigen Receptor (CAR) T cells per kg of recipient bodyweight
  3.0x10^6 Chimeric Antigen Receptor (CAR)+ T cells/kg (weight based dosing) infuse on day 0 and Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 and Fludarabine: 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
- Cohort 1 No Level Assigned - Enrolled But Not Treated; Cohort 2 No Level Assigned - Enrolled But Not Treated: Participants in this group were enrolled but not treated.
Period: Overall Study
Arm/Group | Dose Escalation Cohort 1 Dose Level -1 - 0.15x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 2 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 4 - 9.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 5 - 18x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 2 Dose Level 1 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 2 Dose Level 2 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Cohort 1 No Level Assigned - Enrolled But Not Treated | Cohort 2 No Level Assigned - Enrolled But Not Treated
Started | 0 | 3 | 4 (One participant was enrolled and removed from study with no treatment and was later re-enrolled and treated.) | 8 (One participant was enrolled and removed from study with no treatment and was later re-enrolled and treated.) | 5 | 0 | 3 | 1 | 1 | 1
Completed | 0 | 3 | 3 | 7 | 5 | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Did not receive treatment. | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Enrolled and removed from study with no treatment | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Chemotherapy was started and not finished & no Chimeric Antigen Receptor T-cells were administered. | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 2 participants who had baseline data collected and were enrolled but not treated, is reported here.
Groups:
- Dose Escalation Cohort 1 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg: Participants who have not had an allogeneic hematopoietic stem cell transplant. 0.3x10^6 Chimeric Antigen Receptor (CAR) T cells per kg of recipient bodyweight
  Starting dose: 0.3x10^6 Chimeric Antigen Receptor (CAR)+ T cells/kg (weight based dosing) infuse on day 0 and Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 and Fludarabine: 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
- Dose Escalation Cohort 1 Dose Level 4 - 9.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg: Participants who have not had an allogeneic hematopoietic stem cell transplant. 9.0x10^6 Chimeric Antigen Receptor (CAR) T cells per kg of recipient bodyweight
  9.0x10^6 Chimeric Antigen Receptor (CAR)+ T cells/kg (weight based dosing) infuse on day 0 and Cyclophosphamide: 500 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 and Fludarabine: 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Cohort 1 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 2 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 4 - 9.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 2 Dose Level 1 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 2 Dose Level 2 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Cohort 1 No Level Assigned - Enrolled But Not Treated | Cohort 2 No Level Assigned - Enrolled But Not Treated | Total
Number analyzed (Participants) | 3 | 3 | 7 | 5 | 3 | 1 | 1 | 1 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 7 | 5 | 3 | 1 | 1 | 1 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.13 (6.49) | 42.97 (9.59) | 39.87 (14.8) | 27.94 (13.63) | 28.9 (7.29) | 43.8 (0) | 31.4 (0) | 26.1 (0) | 36.17 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 4 | 1 | 0 | 1 | 1 | 0 | 8
  Male | 3 | 2 | 3 | 4 | 3 | 0 | 0 | 1 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 2 | 3 | 7 | 5 | 2 | 1 | 1 | 1 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 2 | 3 | 6 | 4 | 2 | 1 | 1 | 1 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 7 | 5 | 3 | 1 | 1 | 1 | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Anti-Tumor Necrosis Factor (TNF) Receptor Superfamily Member 8 (CD30) Chimeric Antigen Receptor (CAR) in Participants With Advanced CD30-expressing Lymphomas
Description: Maximum tolerated dose is defined as the dose at which a maximum of 1 of 6 participants has a dose-limiting toxicity (DLT). A DLT is defined as toxicities occurring within 30 days of CAR T-cell infusion. DLT's are Grade 3 or Grade 4 toxicities possibly, probably, or definitely related to either the anti-CD30 CAR T cells or the fludarabine and cyclophosphamide chemotherapy conditioning regimen and lasting more than 7 days. A DLT will only be considered in participants who have received CAR T-cell infusions.
Time Frame: 4-5 weeks after first dose
Measure: Number; unit: million CAR T-cells/kg
Groups:
- All Participants: All participants in Dose Escalation groups Cohort 1 and Cohort 2.
Arm/Group | All Participants
Number analyzed (Participants) | 22
million CAR T-cells/kg | 3

2. Secondary Outcome: Peak Percentage and Persistence at 1 Month of Peripheral Blood Mononuclear Cells (PBMC) That Expressed the Chimeric Antigen Receptor (CAR) T-cells
Description: Peak percentage and the percentage 1 month after infusion of peripheral blood mononuclear cells (PBMC) that expressed the Chimeric Antigen Receptor (CAR) T-cells assessed by polymerase chain reaction (PCR).
Time Frame: From time of infusion until 1 month after infusion
Population: Participants #8, and 23 were not assigned to a dose level since they didn't receive chemo or cells. Participant # 5 first enrolled as #3 did not result in cell infusion and was re-enrolled with a new number for cell infusion. This is the same for #18 who was first enrolled as #16.
Measure: Number; unit: peak percentage
Groups:
- Dose Escalation Cohort 2 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg: Participants who have had an Human Leukocyte Antigen (HLA)-matched sibling or an 8/8-HLA-matched unrelated donor transplant.
  0.3x10^6 Chimeric Antigen Receptor (CAR) T cells per kg of recipient bodyweight
  0.3 x10^6 Chimeric Antigen Receptor (CAR)+ T cells/kg (weight based dosing) infuse on day 0 and Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 and Fludarabine: 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
- Dose Escalation Cohort 2 Dose Level 2 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg: Participants who have had an Human Leukocyte Antigen (HLA)-matched sibling or an 8/8 HLA-matched unrelated donor transplant.
  1.0x10^6 Chimeric Antigen Receptor (CAR) T cells per kg of recipient bodyweight
  1.0x10^6 Chimeric Antigen Receptor (CAR)+ T cells/kg (weight based dosing) infuse on day 0 and Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 and Fludarabine: 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
Arm/Group | Dose Escalation Cohort 1 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 2 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 4 - 9.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 2 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 2 Dose Level 2 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg
Number analyzed (Participants) | 3 | 3 | 7 | 5 | 3 | 1
peak percentage
  Participant #1 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Participant #1 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells | 2.505994998 |  |  |  |  |
  Participant #2 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Participant #2 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells | 1.003513397 |  |  |  |  |
  Participant #4 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Participant #4 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells | 0.257878064 |  |  |  |  |
  Participant #5 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Participant #5 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  | 5.692026394 |  |  |  |
  Participant #6 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Participant #6 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  | 0.066168665 |  |  |  |
  Participant #7 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Participant #7 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  | 0.875579553 |  |  |  |
  Participant #9 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Participant #9 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  |  |  |  | 10.425784436 |
  Participant 10 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Participant 10 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  |  |  |  | 1.173870125 |
  Participant #11 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Participant #11 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  |  | 25.06555951 |  |  |
  Participant #12 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Participant #12 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  |  | 2.061723582 |  |  |
  Participant #13 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Participant #13 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  |  | 0.951813793 |  |  |
  Participant 14 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Participant 14 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  |  | 3.770199852 |  |  |
  Participant #15 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Participant #15 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  |  | 21.6416809 |  |  |
  Participant #17 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Participant #17 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  |  |  |  | 9.701843954 |
  Participant #18 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Participant #18 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  |  | 6.193353177 |  |  |
  Participant #19 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Participant #19 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  |  |  |  |  | NA — As pre-specified by the protocol a participant must receive cells to measure percentage and persistence at 1 month. Participant did not receive CAR T cells, so no CAR T cells could possibly be detected in the blood.
  Participant #20 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Participant #20 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  |  |  | 3.484185735 |  |
  Participant #21 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Participant #21 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  |  |  | 51.30355798 |  |
  Participant #22 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Participant #22 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  |  |  | 29.40752103 |  |
  Participant #24 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Participant #24 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  |  |  | 22.45790377 |  |
  Participant #25 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Participant #25 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  |  |  | 55.04760657 |  |
  Participant #26 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Participant #26 - Peak percentage of CAR+ cells among peripheral blood mononuclear cells |  |  | 25.56426658 |  |  |
  Participant #1 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Participant #1 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion | NA — Below the level of detection. |  |  |  |  |
  Participant #2 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Participant #2 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion | NA — Below the level of detection. |  |  |  |  |
  Participant #4 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Participant #4 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion | NA — Sample not available (participant 4 did not have blood drawn at the 1 month f/u due to not coming to their visit). |  |  |  |  |
  Participant #5 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Participant #5 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  | 0.036582556 |  |  |  |
  Participant #6 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Participant #6 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  | 0.010607229 |  |  |  |
  Participant #7 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Participant #7 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  | 0.002843526 |  |  |  |
  Participant #9 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Participant #9 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  |  |  |  | 0.145937491 |
  #10 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  #10 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  |  |  |  | 0.006382466 |
  Participant #11 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Participant #11 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  |  | NA — Sample not available. Participant 11's CAR T cell blood level could not be determined due to technical problems with the research blood sample. |  |  |
  Participant #12 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Participant #12 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  |  | 2.061723582 |  |  |
  Participant #13 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Participant #13 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  |  | NA — Below the level of detection. |  |  |
  Participant #14 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Participant #14 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  |  | 2.361884069 |  |  |
  Participant #15 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Participant #15 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  |  | 1.584343701 |  |  |
  Participant #17 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Participant #17 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  |  |  |  | 0.09701347 |
  Participant #18 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Participant #18 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  |  | 6.193353177 |  |  |
  Participants #19 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Participants #19 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  |  |  |  |  | NA — As pre-specified by the protocol a participant must receive cells to measure percentage and persistence at 1 month. Participant did not receive CAR T cells, so no CAR T cells could possibly be detected in the blood.
  Participant #20 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Participant #20 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  |  |  | 1.110480727 |  |
  Participant #21 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Participant #21 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  |  |  | 8.51303351 |  |
  Participant #22 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Participant #22 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  |  |  | 11.65873475 |  |
  Participant #24 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Participant #24 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  |  |  | 0.289276145 |  |
  Participant #25 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Participant #25 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  |  |  | 18.33580648 |  |
  Participant #26 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Participant #26 - %CAR+ cells among peripheral blood mononuclear cells 1 month after infusion |  |  | NA — Sample not available (participant 26 did not have blood drawn at the 1 month f/u due to not coming to their visit). |  |  |

3. Secondary Outcome: Number of Participants With Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progression as Their Best Response
Description: Response was measured using the Cheson et al. Revised Response Criteria for Malignant Lymphoma, Journal of Clinical Oncology 2007 and Recommendations for Initial Evaluation, Staging, and Response Assessment of Non-Hodgkin Lymphoma: The Lugano Classification Journal of Clinical Oncology, 2014). Complete Response (CR) is complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. Partial Response (PR) is ≥ 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses. Progressive Disease (PD) ≥ 50% increase from nadir in the sum of the products of at least two lymph nodes, or appearance of a new lesion greater than 1.5 cm in any axis even if other lesions are decreasing in size. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Responses will be assessed as long as the patient is on-study at the following time-points: 1, 2, 3, 4, 6, 9, and 12 months after CAR T-cell infusion. Then responses were assessed every 6 months up until 3 years after CAR T-cell infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort 1 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 2 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 4 - 9.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 2 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 2 Dose Level 2 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg
Number analyzed (Participants) | 3 | 3 | 7 | 5 | 3 | 1
Participants
  Complete Response | 0 | 1 | 0 | 0 | 0 | NA — This participant did not finish chemotherapy and did not receive CAR-T cells so response cannot be assessed.
  Partial Response | 2 | 0 | 3 | 2 | 1 | NA — This participant did not finish chemotherapy and did not receive CAR-T cells so response cannot be assessed.
  Stable Disease | 1 | 2 | 4 | 2 | 2 | NA — This participant did not finish chemotherapy and did not receive CAR-T cells so response cannot be assessed.
  Progressive Disease | 0 | 0 | 0 | 1 | 0 | NA — This participant did not finish chemotherapy and did not receive CAR-T cells so response cannot be assessed.

4. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 11 months and 26 days, 7 months and 10 days, 39 months and 7 days, 17 months and 3 days, 6 months and 15 days, and 1 month and 7 days for each group respectively.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation Cohort 2 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg: Participants who have had an Human Leukocyte Antigen (HLA)-matched sibling or an 8/8-HLA-matched unrelated donor transplant.
  1.0x10^6 Chimeric Antigen Receptor (CAR) T cells per kg of recipient bodyweight
  1.0 x10^6 Chimeric Antigen Receptor (CAR)+ T cells/kg (weight based dosing) infuse on day 0 and Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 and Fludarabine: 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
Arm/Group | Dose Escalation Cohort 1 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 2 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 4 - 9.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 2 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 2 Dose Level 2 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg
Number analyzed (Participants) | 3 | 3 | 7 | 5 | 3 | 1
Participants | 3 | 3 | 7 | 5 | 3 | 1

5. Other Pre Specified Outcome: Number of Participants With a Dose Limiting Toxicity (DLT)
Description: A DLT is defined as toxicities occurring within 30 days of CAR T-cell infusion. DLT's are Grade 3 or Grade 4 toxicities possibly, probably, or definitely related to either the anti-CD30 CAR T cells or the fludarabine and cyclophosphamide chemotherapy conditioning regimen and lasting more than 7 days. A DLT will only be considered in participants who have received CAR T-cell infusions.
Time Frame: 30 days within CAR T-cell infusion
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation Cohort 2 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg: Participants who have had an Human Leukocyte Antigen (HLA)-matched sibling or an 8/8-HLA-matched unrelated donor transplant.
  1.0x10^6 Chimeric Antigen Receptor (CAR) T cells per kg of recipient bodyweight
  1.0x10^6 Chimeric Antigen Receptor (CAR)+ T cells/kg (weight based dosing) infuse on day 0 and Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 and Fludarabine: 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
Arm/Group | Dose Escalation Cohort 1 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 2 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 4 - 9.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 2 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 2 Dose Level 2 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg
Number analyzed (Participants) | 3 | 3 | 7 | 5 | 3 | 1
Participants
  Grade 3 possibly related | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 probably related | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 definitely related | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 possibly related | 0 | 0 | 0 | 1 | 0 | 0
  Grade 4 probably related | 0 | 0 | 0 | 1 | 0 | 0
  Grade 4 definitely related | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 11 months and 26 days, 7 months and 10 days, 39 months and 7 days, 17 months and 3 days, 6 months and 15 days, and 1 month and 7 days for each group respectively.
Arm/Group | Dose Escalation Cohort 1 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 2 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 1 Dose Level 4 - 9.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 2 Dose Level 1 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg | Dose Escalation Cohort 2 Dose Level 2 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/7 | 0/5 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 5/7 | 3/5 | 0/3 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 7/7 | 5/5 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Cohort 1 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg (N=3) | Dose Escalation Cohort 1 Dose Level 2 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg (N=3) | Dose Escalation Cohort 1 Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg (N=7) | Dose Escalation Cohort 1 Dose Level 4 - 9.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg (N=5) | Dose Escalation Cohort 2 Dose Level 1 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg (N=3) | Dose Escalation Cohort 2 Dose Level 2 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg (N=1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, EBV positive B-cell (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Cohort 1 Dose Level 1 - 0.3x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg (N=3) | Dose Escalation Cohort 1 Dose Level 2 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg (N=3) | Dose Escalation Cohort 1 Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg (N=7) | Dose Escalation Cohort 1 Dose Level 4 - 9.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg (N=5) | Dose Escalation Cohort 2 Dose Level 1 - 1.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg (N=3) | Dose Escalation Cohort 2 Dose Level 2 - 3.0x10^6 Chimeric Antigen Receptor (CAR) T Cells Per kg (N=1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (3) | 1 (8) | 3 (21) | 4 (28) | 1 (5) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 2 (7) | 1 (2) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epstein-Barr virus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 2 (2) | 1 (1)
Fever (General disorders) | 1 (2) | 1 (1) | 3 (4) | 3 (16) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, Specify (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — prior Neupogen injection site is erythematous and warm with a darkened center.
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (17) | 2 (5) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (10) | 2 (4) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 1 (8) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 7 (19) | 3 (18) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (3) | 5 (9) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymph node pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (12) | 3 (13) | 7 (40) | 5 (40) | 3 (22) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Nervous system disorders - Other, Numbness in medial side of left forearm (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (16) | 3 (25) | 7 (39) | 5 (34) | 3 (14) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (7) | 5 (24) | 2 (20) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (5) | 4 (7) | 1 (2) | 0 (0)
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, Burning at the end of urination with cramping (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shingles (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (2) | 3 (4) | 5 (11) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 3 (22) | 3 (15) | 7 (43) | 5 (51) | 2 (16) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT03049449/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT03049449/ICF_001.pdf